CLINICAL TRIAL: NCT06152497
Title: The Role of Histamine in Muscle Protein Synthesis Following Chronic Resistance Training
Brief Title: The Role of Histamine in Muscle Protein Synthesis Following Resistance Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MPSH - ONZ-2023-0027
Record Dates: First submitted 2022-12-20; First posted 2023-11-30 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Histamine
MeSH Terms: interventions — fexofenadine; Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel groups
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1: Placebo (Placebo Comparator): Lactose
  Interventions: Drug: Placebo; Behavioral: Resistance training
- H1 blockade: Telfast (180mg Fexofenadine) (Experimental): H1: Telfast (180mg Fexofenadine)
  Interventions: Drug: H1 blockade: Telfast: 180mg Fexofenadine; Behavioral: Resistance training

INTERVENTIONS:
Drug: Placebo — Oral placebo
  Arms: 1: Placebo
Drug: H1 blockade: Telfast: 180mg Fexofenadine — H1 blockade: oral blockade with 180mg Fexofenadine
  Arms: H1 blockade: Telfast (180mg Fexofenadine)
Behavioral: Resistance training — Resistance training: lower body exercise

SUMMARY:
Blocking histamine H1/H2 receptors blunts chronic endurance training adaptations. The current study addresses the following research question: "What is the influence of histamine H1 signaling on training adaptations following ten weeks of resistance training in human skeletal muscle." Results from this study will yield more insights into the molecular mechanisms of adaptations to exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-45 years
* Not to medium physically active

Exclusion Criteria:

* Smoking
* Chronic disease
* High blood pressure
* Supplement or medication intake
* Seasonal allergies
* Vegetarian / vegan
* Resistance trained

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle volume | Before and after the 10 weeks of resistance training
  Change in muscle volume
Maximal dynamic strength of leg press, bench press, bicep curl and leg curl | Before and after the 10 weeks of resistance training
  Change in maximal dynamic strength of leg press, bench press, bicep curl and leg curl
Muscle fiber hypertrophy in muscle biopsies | Before and after the 10 weeks of resistance training
  Change in muscle fiber hypertrophy in muscle biopsies
Matsuda index, to estimate whole body glucose metabolism, will be calculated using an oral glucose tolerance test (OGTT: concentration of glucose and insulin in the blood will be measured before and after drinking 75g glucose) | Before and after the 10 weeks of resistance training
  Change in Matsuda index, to estimate whole body glucose metabolism, will be calculated using an oral glucose tolerance test (OGTT: concentration of glucose and insulin in the blood will be measured before and after drinking 75g glucose)
Vascular function measured with a single passive leg movement (sPLM: change in femoral blood flow measured with Doppler ultrasound before and after one passive flexion/extension of the leg) | Before and after the 10 weeks of resistance training
  Change in vascular function with a single passive leg movement (sPLM: change in femoral blood flow measured with Doppler ultrasound before and after one passive flexion/extension of the leg)

SECONDARY OUTCOMES:
Blood pressure (systolic and diastolic) | Before and after the 10 weeks of resistance training
  Chance in Blood pressure (systolic and diastolic)
Resting heart rate | Before and after the 10 weeks of resistance training
  Chance in Resting heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Wim Derave, Professor, Principal Investigator — University Ghent
Locations (1):
- Department of movement and sports sciences, Ghent University, Belgium, Ghent, Oost-Vlaanderen, Belgium